CLINICAL TRIAL: NCT06835842
Title: Effect of Rib Mobilization on Weaning Parameters From Mechanical Ventilator in Patients With Pneumonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Gaber, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT REC/012/005446
Record Dates: First submitted 2025-02-09; First posted 2025-02-19 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rib mobilization technique and routine chest physiotherapy group (Experimental): 1.rib mobilization technique and routine chest physio therapy group: the patients will receive rib mobilization technique in addition to their medical treatment and routine chest physiotherapy for at least 30 minutes once daily for ten consecutive days
  Interventions: Other: rib mobilization technique; Other: routine chest physiotherapy
- routine chest physiotherapy group (Active Comparator): routine chest physiotherapy group : the patients in this group will receive routine chest physical therapy for at least 30 minutes once daily for 10 consecutive days
  Interventions: Other: routine chest physiotherapy

INTERVENTIONS:
Other: rib mobilization technique — rib mobilization technique The patient in experimental group will be relaxed in semi- fowler position while connected to mechanical ventilator, therapist will seat at the patient "side, his fingers pads are placed at the position of the patient's rib angles , pulling upward and the lateral position the position is held while wait for the soft tissues to release this take from 15 seconds .Release of the diaphragm through manual contact with hypothenar region of therapist thumb inferior laterally xiphoid process and rest along Antero lateral costal margin below rib7 during exhalation the therapist thumb give pressure posteriorly repeat this steps for 3 to5 respiratory cycle • routine chest physiotherapy percussion on chest wall its frequency should be 3-7 beats per sec. vibration applying a light pressure with hand on affected segment for about 5 min modified postural drainage R. and L. side. U&L limb passive ex. for R.10 x3 set
  .this program for 30 minutes once daily for ten days
  Arms: rib mobilization technique and routine chest physiotherapy group
Other: routine chest physiotherapy — routine chest physiotherapy the patient will be laid in half supine position connected to a ventilator applying
  * percussion on chest wall its frequency should be 3-7 beats per second or 180-420 beats per minute
  * vibration applying a light pressure with flattened hand on affected segment for about 5 minutes
  * modified postural drainage (right and left sidling 10 min for each side
  * upper and lower limb exercise for 4 limbs (3 sets and each set has 10 repetition
  * this program for 30 minutes once daily
  * for 10 consecutive days

SUMMARY:
this study will be conducted to distinguish between effect of rib mobilization and routine chest physiotherapy on weaning parameters from mechanical ventilator in patients with pneumonia •

HYPOTHESES:

It will be hypothesized that there may be significant effect of rib mobilization on weaning parameters from mechanical ventilator in patients with pneumonia.

RESEARCH QUESTION:

Does rib mobilization have an effect on weaning parameters from mechanical ventilator in patients with pneumonia? measuring weaning parameters: on screen of mechanical ventilator : measuring respiratory rate, Tidal volume (TV), FiO2.

* Arterial blood gases (ABG) analyzer machine ABG is recorded daily (PH- PaO2 - PaCO2)
* Length of ICU stay: calculated by (admission date - discharge date
* Weaning success rate

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) represents a significant sub-set of (HAP) remains the most frequent intensive care unit (ICU)-acquired infection its incidence ranges from 9% to 27% of ventilated patients ,VAP is associated with an increased length of stay, mortality and health care costs, Pneumonia can result in chest wall stiffness, decreased mobility, limiting the range of motion during breathing and decreased lung compliance and impaired respiratory function , Rib mobilization: is an articular , non-invasive, passive technique that can be useful with acutely ill, hospitalized patients emphasizes the placement of a repetitive force to increase the range of motion of the posterior rib articulations and chest wall , lessening somatic dysfunction of the spine, stretches myofascial structures and improve respiratory mechanics So, this study will be conducted to distinguish between effect of rib mobilization and routine chest physiotherapy on weaning parameters among intubated pneumonic patients on mechanical vent.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age ranged from 40- 50 years old from both genders.
2. Diagnosed with pneumonia and need invasive mechanical ventilation support.
3. Stable oxygen saturation (SpO2 more than 85, (FiO2) 0.6 or less, PEEP less than 10 Cm H2O).
4. mean arterial pressure > 75 mmHg and urine output > 1 mL/kg/h;
5. Patients with Glasgow coma scale (GCS) > 8T
6. Unconscious and semi-conscious patients. -

Exclusion Criteria:

1. Unstable hemodynamics
2. Unstable neurological problems e.g. (epileptic seizures -hyperthermia).
3. Unstable chest wall e.g. (multiple rib or vertebral fractures)
4. Increase intracranial pressure (>20 mmHg for >5 min).
5. Undrained pneumothorax, recent pulmonary surgery

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Arterial blood gases | at least 10 consecutive days
  • Arterial blood gases (ABG): (PH -PaO2 - PaCO2)
  • PaO2/FiO2 ratio (P/F): One element of predicting successful weaning from mechanical ventilation is PaO2/FiO2 > 200
Respiratory rate (RR) | at least 10 consecutive days
  It will be measured using a mechanical ventilator.
Tidal volume (TV) | at least 10 consecutive days
  It will be measured using a mechanical ventilator.

SECONDARY OUTCOMES:
Length of hospital stay | at least 10 consecutive days
  ;• Length of stay in intensive care unite can be defined as the number of days that an in-patient will remain in ICU during a single admission event, is calculated by subtracting the admission date (ADATE) from the discharge date (DDATE)

CONTACTS AND LOCATIONS:
Overall Officials: Azza Abd El Aziz Abd El Hady, professor, Study Chair — Cairo University; Mohammed Abd Hakim El-Nadi, professor, Study Director — Cairo University
Locations (1):
- El Galaa Military Hospital, Cairo, Egypt